CLINICAL TRIAL: NCT00170105
Title: Posturing Effects on Perception of Time and Perceptions of the Provider-Patient Interaction in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Annie T. Sadosty, M.D., Mayo Clinic
Other Study IDs: 1487-05
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Age 18 years or older; No cognitive impairment or altered mental status; Stable; No aphasia; English-speaking

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study Objective:

* To examine the perceptions of time spent at the bedside; perceptions of bedside manner; and patient perceptions of the provider-patient interaction offered by emergency providers when they sit versus when they stand during the initial evaluation.

This project is clinically relevant research different from prior Emergency Department (ED) satisfaction studies since this study will contribute information about factors that could increase patient satisfaction with his/her provider in the ED setting. This research may guide specific guidelines for quality improvement efforts. The investigators hypothesize that patients will perceive that the emergency providers are at the bedside longer, demonstrate better bedside manner, and have better provider-patient interactions when they sit versus when they stand. Additionally, the investigators hypothesize that providers who sit will perceive that they are at the bedside longer than those who stand for the same period of time.

Methods: A convenience sample of adult patients will complete a 5-item questionnaire concerning the perceived time spent with the emergency provider and the qualities of the provider-patient interaction. Emergency providers will be randomly assigned to either sit or stand during the initial evaluation. The providers will complete a 4-item questionnaire. These data will be compared to the actual time spent in the evaluation, measured in seconds, using a stopwatch. These data, combined with demographic data obtained from the patient chart, will be analyzed to examine whether there are statistically significant differences in patient perceptions and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* The subject population represents a convenience sample of patients 18 years and older who give consent.
* All English speaking individuals with adequate health status and cognitive function to communicate answers to the investigator.
* There are no foreseen reasons to exclude pregnant women as they are not likely to be vulnerable in this study.

Exclusion Criteria:

* Unstable patients and patients seen in the critical care area will be excluded from study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: •- The subject population represents a convenience sample of patients 18 years and older who give consent.
  * All English speaking individuals with adequate health status and cognitive function to communicate answers to the investigator.
  * There are no foreseen reasons to exclude pregnant women as they are not likely to be vulnerable in this study.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2005-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie T. Sadosty, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States